CLINICAL TRIAL: NCT03579797
Title: Shanghai Eye Disease Prevention and Treatment Center
Brief Title: Shanghai Diabetic Eye Study in Diabetics
Acronym: SDES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Principal Investigator, Jiannan Huang, Shanghai Eye Disease Prevention and Treatment Center, Shanghai Eye Disease Prevention and Treatment Center
Other Study IDs: YFZX2018005
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Eye Diseases; Diabetic Retinopathy
Keywords: diabetic eye diseases; diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Mass Screening; Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The morning urine and the fasting blood will be collected for testing, including blood routine, blood glucose, glycosylated hemoglobin, liver and kidney function, blood lipid, urine microalbumin, urine albumin/creatinine ratio etc.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Screening, referral, follow-up and health management — Field screening, remote diagnosis, comprehensive assessment, referral, and eye health management of diabetics were the main study processes. The community health service centers (CHSC) are responsible for the field screening. The designated medical institutions (DMI) of each district are responsible for the remote diagnosis and comprehensive assessment of diabetic eye diseases, especially diabetic retinopathy (DR), based on comprehensive evaluation through the remote reading system (RRS) and Shanghai eye health information service system (SEHISS). The staff of CHSC urged the referral objects promptly for further diagnosis and treatment in DMI. According to the diagnosis after clinically confirmed, all the study participants will be recommended appropriate eye health management.

SUMMARY:
The purpose of the Shanghai Diabetic Eye Study (SDES) was to guide and regulate eye health screening of two hundred thousand people with diabetes in the communities in 16 districts in Shanghai, build up the ranks with the general practitioner as the backbone combined, and provide comprehensive, continuous, and dynamic information service to diabetic eye disease health management. We expect to form a "screening, finding, referral, follow-up and health management" diabetic eye disease working mode, integrate medical care and precaution closely, promote the classified management and referral, reduce the prevalence rate of diabetic eye disease, blindness and visual impairment of DR, and improve diabetics consciousness of eye health maintenance. At the same time, we will also improve the device configuration of eye health screening and relevant personnel training mechanism in the community health service centers, thus upgrading the level of eye disease prevention and treatment in Shanghai.

DETAILED DESCRIPTION:
Community-based cross-sectional samples of the archives management of adults with diabetes aged 35 years and above in 241 community health service centers (CHSC) in 16 districts in Shanghai, were obtained through proportional sampling (32%). Field screening, remote diagnosis, comprehensive assessment, referral, and eye health management of diabetics were the main study processes. Field screening mainly included visual acuity assessment, autorefraction examination, and non-mydriatic fundus photography. The designated medical institutions (DMI) of each district are responsible for the remote diagnosis and comprehensive assessment of diabetic eye diseases, especially diabetic retinopathy (DR), based on comprehensive evaluation of eye and general condition through the remote reading system (RRS) and Shanghai eye health information service system (SEHISS). The staff of CHSC urged the referral objects promptly for further diagnosis and treatment in DMI. According to the diagnosis after clinically confirmed, all the study participants will be recommended appropriate eye health management

ELIGIBILITY:
Inclusion Criteria:

* The target population included the adults with diabetes aged 35 years and above under archives management, residing in Shanghai.

Exclusion Criteria:

* <35 years old;
* Diabetics should not be able to move freely, clear-thinking and considered possible to cooperatively complete the ophthalmic examinations.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sampling was carried out in a proportional sampling plan that each diabetic under the archives management aged 35 years and above, residing in Shanghai.
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetic retinopathy | December 31, 2018
  Prevalence of DR and diabetic macular edema. The DR grades are according to the well-accepted"International Clinical Diabetic Retinopathy and Diabetic Macular Edema Disease Severity Scale".
Diabetic eye diseases | December 31, 2018
  Prevalence of eye diseases due to diabetes.
Visual impairment | December 31, 2018
  Visual impairment was present if best corrected visual acuity <20/25
Glycosylated hemoglobin | December 31, 2018
  This test measure the average blood sugar control for the previous three months or so.
Diabetics adherence to Diabetic Eye Diseases Study | December 31, 2018
  Predicting adherence in the research were obtained by Questionnaire for the study participants.
Diabetics satisfaction for the SDES | December 31, 2018
  Diabetics satisfaction for the screening study，the community health service centers (CHSC)，and the designated medical institutions were obtained by Questionnaire for the study participants.
Referral compliance | December 31, 2018
  Referral compliance of diabetics were obtained by Questionnaire and Shanghai eye health information service system for the study participants.
Human resources and ophthalmic equipment resources | December 31, 2018
  Compared to human resources and ophthalmic equipment resources in the community health service centers (CHSC)，and the designated medical institutions before and after the SDES by Questionnaire.
Eye health management | December 31, 2018
  All the study participants will be recommended appropriate eye health management.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zou, MD，PhD, Study Chair — Shanghai Eye Disease Prevention and Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Jingan, China